CLINICAL TRIAL: NCT00617721
Title: Defect in Cell Stimulation and Unexplained hemorrhagesMarkers Related to Membrane Remodelling in the Prognosis Scott-like Syndormes
Brief Title: Markers of Defective Membrane Remodelling in Scott-like Syndromes
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Louis Pasteur University, Strasbourg (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Aventis, Génopôle d'Evry. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3930
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Unexplained Isolated Provoked Hemorrhages; Familial Bleeding Disorder; Scott Syndrome
Keywords: Defective gene(s) in plasma membrane remodelling.; Scott syndrome,; Reduced prothrombin consumption,; Circulating biomakers of scott syndrome
MeSH Terms: conditions — Scott Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, white cells, DNA (when the family is informative)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with unexplained bleeding disorder
  Interventions: Other: Blood withdrawal
- 2: healthy volunteers
  Interventions: Other: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal — Observational study. Limited blood withdrawal. Any other intervention will be determined by the patient's clinical status.

SUMMARY:
Purpose: Identification of the gene(s) involved in plasma membrane remodelling. Identification of the circulating markers affected by the defective membrane remodelling in a collection of families with unexplained provoked hemorrhages and evaluation of their prognosis value in the assessment of the hemostatic cellular response.Hypothesis: Scott syndrome is rare a familial disorder characterized by provoked haemorrages in homozygous-type patients due to isolated membrane remodelling deficiency. Membrane remodelling is necessary for cellular hemostatic responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unexplained provoked hemorrhages (surgery, tooth extraction, birth …), and associated with reduced prothrombin consomption (residual prothrombine in serum > à 5%).
* Family members of the patients defined above, with or without unexplained hemorrhages (symptomatic or not).
* Patient's approval based on detailed information given by the pratician

Exclusion Criteria:

* Patients with primary hemostasis defect or defective blood coagulation factor(s) possibly explaining the bleeding disorder.
* Anémia,
* patients known to be affected by Factor V New York .
* Patients enrolled in a previous clinical study, the exclusion period of which is not yet completed. - Collaboration to the study rejected by the patient
* Patients that are not registered for medical care social insurance.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unexplained bleeding disorder
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: Lélia GRUNEBAUM, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (5):
- France (4):
  - Hôpital Antoine Béclère, Service d'Hématologie Biologique, Clamart
  - Laboratoire d'Hémostase et d'Immunologie, Centre Hospitalier, Le Mans
  - Laboratoire d'Hématologie, Hôpital Robert Debré, Reims
  - Laboratoire d'Hématologie, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
- Service d'Hématologie Biologique, Hôpital Pierre Zobda Quitman, Fort-de-France, Martinique